CLINICAL TRIAL: NCT04855591
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose-Escalation Study to Evaluate the Safety, Tolerability, PK, PD and Immunogenicity of Single Subcutaneous Administered SHR-1703 in Healthy Caucasian Subjects
Brief Title: A Trial of SHR-1703 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of the clinical development plan for this product globally
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1703-104-AUS
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR-1703 Dose Level 1 (Experimental): Dose level 1 SHR-1703
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703 Dose Level 2 (Experimental): Dose level 2 SHR-1703
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703 Dose Level 3 (Experimental): Dose level 3 SHR-1703
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703 Dose Level 4 (optional) (Experimental): Dose level 4 SHR-1703 Additional dose escalations, as determined by the SMC depend on PK and safety data review
  Interventions: Drug: SHR-1703; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1703 — SHR-1703 will be administered subcutaneously
Drug: Placebo — Placebo of SHR-1703 will be administered subcutaneously

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single dose escalation phase 1 study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics pharmacodynamics and immunogenicity of subcutaneous administered SHR-1703 in healthy subjects.

DETAILED DESCRIPTION:
The study will consist of one dose esclation part with a total of 3 dose levels. The Subjects will be randomized to receive SHR-1703 as reflected by the guiding principle for the dose esclation/expansion phase. Each dose group includes a screening period, a baseline period, an observational period, and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian subjects, male and female, 18 to 55 years of age, inclusive;
2. Body weight ≥45 kg (Both male and female), body mass index (BMI) between ≥19.0 and ≤29.9 kg/m2, inclusive;
3. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry and coagulation function) and ECG at the investigator's discretion during screening and baseline.
4. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods and have no plan to have a child from signing the consent form to 30-days after last scheduled follow-up visit.

Exclusion Criteria:

1. Known history or suspected of being allergic to the study drug.
2. Positive hepatitis B virus (HBsAg), hepatitis C virus (HCV-Ab), human immunodeficiency virus (HIV-Ab) at screening.
3. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening or within 5 half-lives of any drugs during screening visit, or in the follow-up period of a clinical study whichever is longer
4. Use of any medicine within 4-weeks prior to the IP administration
5. Blood donation or loss of more than 400 mL of blood within 1 month of screening; or received blood transfusion within 2 months before screening.
6. Live (attenuated) vaccination within 1 month before screening or plan to be vaccinated
7. Severe injuries or major surgeries within 6 months before screening or plan to do surgeries during the trial
8. Patients with known or suspected parasitic infection within 6 months before screening
9. Either ALT, AST, ALP, GGT or total bilirubin level exceeds upper limit of normal range (ULN) at screening or baseline visits (confirmed by a single repeat, as per investigator's judgment)
10. More than 5 cigarettes daily (or products with equivalent amount of nicotine) for 3 months prior to screening.
11. History of alcohol abuse within 3 months prior to the IP administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 34 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 34 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1703 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 34 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1703 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 34 weeks)
  Time to Cmax of SHR-1703
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 34 weeks)
  Maximum observed concentration of SHR-1703
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 34 weeks)
  Apparent clearance of SHR-1703
Pharmacokinetics-Vz/F | Start of Treatment to end of study (approximately 34 weeks)
  Apparent volume of distribution during terminal phase of SHR-1703
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 34 weeks)
  Terminal elimination half-life of SHR-1703
Pharmacodynamics-Eosinophils | Start of Treatment to end of study (approximately 34 weeks)
  Absolute eosinophils account and change from baseline in percentage
Anti-drug-antibody | Start of Treatment to week 22 after IP administration
  The percentage of subjects with positive ADA titers over time for SHR-1703

CONTACTS AND LOCATIONS:
Overall Officials: Dr Richard Friend, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No